CLINICAL TRIAL: NCT00762229
Title: Prospective Evaluation of LDL Levels in Patients Converted From Zetia (Ezetimibe)10 mg to 5 mg
Brief Title: Evaluation of LDL Cholesterol in Patients Switched From 10 to 5 Milligrams of Zetia (Ezetimibe)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bronx VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Lawrence Baruch, Staff physician, Bronx VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: VA---19-07-051
Record Dates: First submitted 2008-09-29; First posted 2008-09-30 (Estimated); Results first posted 2013-06-14 (Estimated); Last update posted 2013-06-14 (Estimated); Status verified 2013-06

CONDITIONS: Hypercholesterolemia
Keywords: Cholesterol; Ezetimibe
MeSH Terms: conditions — Hypercholesterolemia | interventions — Ezetimibe

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ezetimibe 10 mg (Active Comparator): A whole ezetimibe 10 mg tablet
  Interventions: Drug: Ezetimibe 10 mg
- Ezetimibe 5 mg (Experimental): Ezetimibe 5 mg, "formulated" by splitting a 10 mg ezetimibe tablet in half
  Interventions: Drug: Ezetimibe 5 mg

INTERVENTIONS:
Drug: Ezetimibe 10 mg — Ezetimibe 10 mg daily for 4 weeks
  Other Names: Zetia
  Arms: Ezetimibe 10 mg
Drug: Ezetimibe 5 mg — Ezetimibe 5 mg daily for 4 weeks, "formulated" as a 10 mg tablet split in half
  Other Names: Zetia
  Arms: Ezetimibe 5 mg

SUMMARY:
The purpose of this study is to compare the effect on LDL cholesterol levels of converting patients who are receiving the cholesterol absorption inhibitor Zetia at a dose of 10 milligrams to 5 milligrams, when prescribed as a split 10 milligram tablet.

ELIGIBILITY:
Inclusion Criteria:

* Subjects receiving ezetimibe 10 mg
* Subjects who have demonstrated compliance with ezetimibe as evidenced by the following Proportions of Days Covered patterns (which represent a PDC of more than 75%):

  * 90 day prescriptions: Filled a ezetimibe prescription within the previous 4 months
  * 60 day prescriptions: Filled a ezetimibe prescription within the previous 2.5 months
  * 30 day prescriptions: Filled a ezetimibe prescription within the previous 1.5 months
* Patients willing and able to provide signed informed consent

Exclusion Criteria:

* Patients not receiving ezetimibe
* Patients receiving ezetimibe 5 milligrams
* Patients with a history of being titrated from ezetimibe 5 to 10 mg. Stroke,TIA, myocardial infarction, unstable angina, percutaneous coronary intervention, coronary artery bypass surgery, or major surgery within the 3 months
* Cancer undergoing active treatment
* Participation in any clinical study within the last 30 days
* Drug addiction or alcohol abuse within the past 6 months
* Patients unwilling or unable to provide informed consent
* Patients with poor compliance
* Women of childbearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2007-07; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Baruch, MD, Principal Investigator — Bronx VA Medical Center
Locations (1):
- Bronx VA Medical Center, The Bronx, New York, United States

REFERENCES:
- [Result] Baruch L, Agarwal S, Gupta B, Haynos A, Eng C. Effect on serum lipid levels of switching dose of ezetimibe from 10 to 5 mg. Am J Cardiol. 2009 Jun 1;103(11):1568-71. doi: 10.1016/j.amjcard.2009.01.365. Epub 2009 Apr 22. PMID 19463517

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from themedical, cardiology and lipid clinics from Spetember 2007 through April 2008.
Pre-assignment Details: The drug was prescribed once daily. No patients were excluded after randomization
Groups:
- Ezetimibe 5 mg: Ezetimibe 5 mg,
Period: Overall Study
Arm/Group | Ezetimibe 10 mg | Ezetimibe 5 mg
Started | 15 | 24
Completed | 14 | 22
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — did not recveive intervention | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ezetimibe 10 mg | Ezetimibe 5 mg | Total
Number analyzed (Participants) | 15 | 24 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 9 | 19
  >=65 years | 5 | 15 | 20
Age Continuous [Mean (Standard Deviation); unit: years] | 69 (9.2) | 72 (10.1) | 70.5 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 15 | 23 | 38
Region of Enrollment [Number; unit: participants]
  United States | 15 | 24 | 39

OUTCOME MEASURES:

1. Primary Outcome: LDL Cholesterol
Description: LDL cholesterol
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Ezetimibe 10 mg | Ezetimibe 5 mg
Number analyzed (Participants) | 14 | 22
mg/dL | 103 (24) | 97 (38)

2. Secondary Outcome: Total Cholesterol
Description: Total cholesterol fasting
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Ezetimibe 10 mg | Ezetimibe 5 mg
Number analyzed (Participants) | 14 | 22
mg/dL | 180 (35) | 167 (48)

ADVERSE EVENTS:
Description: The saftey population includes all participants who received at least one dose of study drug and who were not lost to follow up.
Arm/Group | Ezetimibe 10 mg | Ezetimibe 5 mg
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/23
Other Adverse Events (participants affected / at risk) | 0/15 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No